CLINICAL TRIAL: NCT02270606
Title: Phase I Study of Neoadjuvant Short Course Radiotherapy Concurrent With Infusional 5-Fluorouracil for the Treatment of Locally Advanced Rectal Cancer
Brief Title: Phase I Study of Neoadjuvant Radiotherapy With 5-Fluorouracil for Rectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-14-10491; NCI-2014-02089 (Registry Identifier: NCI CTRP); P30CA016059 (NIH)
Record Dates: First submitted 2014-10-16; First posted 2014-10-21 (Estimated); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Mucinous Adenocarcinoma of the Rectum; Recurrent Rectal Cancer; Signet Ring Adenocarcinoma of the Rectum; Rectal Adenocarcinoma; Stage IIA Rectal Cancer; Stage IIB Rectal Cancer; Stage IIC Rectal Cancer; Stage IIIA Rectal Cancer; Stage IIIB Rectal Cancer; Stage IIIC Rectal Cancer
Keywords: Rectum
MeSH Terms: conditions — Rectal Neoplasms | interventions — Radiotherapy, Intensity-Modulated; Fluorouracil; dehydroftorafur; Oxaliplatin; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment(IMRT,fluorouracil,chemotherapy,surgery) (Experimental): CHEMORADIATION:Patients undergo Intensity Modulated Radiation Therapy (IMRT) once a day over 5 days for total of 5 fractions and concurrently receive fluorouracil IV continuously over 96 hours.
  PREOPERATIVE CHEMOTHERAPY:Within 2 weeks of completing chemoradiation, patients receive oxaliplatin IV over 2 hours, leucovorin calcium IV over 2 hours, and fluorouracil IV as a push followed by IV continuously over 46 hours on day 1.Treatment repeats every 14 days for 4 courses in absence of disease progression or unacceptable toxicity.
  SURGERY:Within 4-8 weeks of completing preoperative chemotherapy, patients undergo total mesorectal excision as therapeutic conventional surgery.
  POSTOPERATIVE CHEMOTHERAPY:Within 4-8 weeks after surgery, patients receive oxaliplatin, leucovorin calcium, and fluorouracil(preoperative chemotherapy).Treatment repeats every 14 days for 6 courses in absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: intensity-modulated radiation therapy; Drug: fluorouracil; Drug: oxaliplatin; Drug: leucovorin calcium; Procedure: therapeutic conventional surgery

INTERVENTIONS:
Radiation: intensity-modulated radiation therapy — Undergo IMRT
  Other Names: IMRT
Drug: fluorouracil — Given IV
  Other Names: 19893; 2,4-Dioxo-5-fluoropyrimidine,; 5-Fluoro-2,4(1H,3H)-pyrimidinedione,; Actino-Hermal, Adrucil; Arumel
Drug: oxaliplatin — Given IV
  Other Names: 1-OHP, 63121-00-6, [(1R,-2R)-1,2-cyclohexanediamine-N,N']; diaminocyclohexane; oxalatoplatinum; Dacotin; Dacplat
Drug: leucovorin calcium — Given IV
  Other Names: 1492-18-8, 27275, 3590, 4292,; 5-formyl tetrahydrofolate; Adinepar; calcium (6S)-folinate; Calcifolin
Procedure: therapeutic conventional surgery — Undergo total mesorectal excision

SUMMARY:
This phase I trial studies the side effects and best dose of fluorouracil when given together with radiation therapy followed by combination chemotherapy before and after surgery in treating patients with rectal cancer that has spread from where it started to nearby tissue or lymph nodes. Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. Drugs used in chemotherapy, such as fluorouracil, leucovorin calcium, and oxaliplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving more than one drug (combination chemotherapy) before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Giving additional combination chemotherapy after surgery may kill any remaining tumor cells. Giving radiation therapy and fluorouracil followed by combination chemotherapy before and after surgery may be a better treatment for rectal cancer.

DETAILED DESCRIPTION:
OUTLINE: This is a dose-escalation study of fluorouracil.

CHEMORADIATION: Patients undergo intensity-modulated radiation therapy (IMRT) once daily (QD) over 5 days for a total of 5 fractions and concurrently receive fluorouracil intravenously (IV) continuously over 96 hours.

PREOPERATIVE CHEMOTHERAPY: Within 2 weeks of completing chemoradiation, patients receive oxaliplatin IV over 2 hours, leucovorin calcium IV over 2 hours, and fluorouracil IV as a push followed by IV continuously over 46 hours on day 1. Treatment repeats every 14 days for 4 courses in the absence of disease progression or unacceptable toxicity.

SURGERY: Within 4-8 weeks of completing preoperative chemotherapy, patients undergo total mesorectal excision.

POSTOPERATIVE CHEMOTHERAPY: Within 4-8 weeks after surgery, patients receive oxaliplatin, leucovorin calcium, and fluorouracil as in preoperative chemotherapy. Treatment repeats every 14 days for 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 1 year or until removal from the study or death, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically proven diagnosis of adenocarcinoma of the rectum (located below the peritoneal reflection or begins within 15 cm of the anal verge on flexible endoscopy) within 90 days of registration; diagnosis of rectal adenocarcinoma must be obtained by biopsy technique that does not completely excise the lesion (eg, fine needle aspiration, core needle biopsy)
* Clinically determined to be clinically staged (American Joint Committee on Cancer (AJCC) 7th edition [ed.]) T3-4 N0 M0 or T any N1-2 M0 based upon the following minimum diagnostic workup within 90 days prior to registration:

  * Colonoscopy
  * History/physical examination (including medication history screen for contraindications)
  * Contrast-enhanced imaging of the abdomen and pelvis either by computed tomography (CT), magnetic resonance imaging (MRI), or whole body positron emission tomography (PET)-CT (preferred)
  * Chest x-ray (or CT) of the chest to exclude distant metastases (except for those who have had whole body PET-CT per above bullet point)
  * Transrectal ultrasound (TRUS) or MRI for T staging
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1
* Absolute neutrophil count (ANC) >= 1,800 cells/mm^3
* Platelets >= 100,000 cells/mm^3
* Hemoglobin >= 8.0 g/dL (note: the use of transfusion or other intervention to achieve hemoglobin [Hgb] >= 8.0 g/dL is acceptable)
* Aspartate aminotransferase (AST) < 2.5 x upper limit of normal (ULN)
* Alkaline phosphatase < 2.5 x ULN
* Bilirubin =< 1.5 ULN
* Calculated creatinine clearance (CrCl) > 50 mL/min using Cockcroft-Gault formula
* Must be deemed a candidate for curative resection by the surgical oncologist who will be performing the operation
* Must provide study-specific informed consent prior to study entry
* Must have a negative serum pregnancy test

Exclusion Criteria:

* Prior radiotherapy to the region of the body that would result in overlap of RT fields with the current protocol treatment
* Severe, active comorbidity, defined as follows:

  * Unstable angina and/or congestive heart failure requiring hospitalization within the last 12 months
  * Transmural myocardial infarction within the last 6 months
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
  * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy within 30 days prior to registration
  * Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects
  * Acquired immune deficiency syndrome (AIDS) based upon current Centers for Disease Control and Prevention (CDC) definition; note, however, that human immunodeficiency virus (HIV) testing is not required for entry into this protocol
  * Evidence of uncontrolled seizures, central nervous system disorders, or psychiatric disability judged by the investigator to be clinically significant, precluding informed consent, or interfering with compliance of treatment protocol or follow up
  * Known, existing uncontrolled coagulopathy; subjects on therapeutic anticoagulation may be enrolled provided that they have been clinically stable on anti-coagulation for at least 2 weeks
  * Major surgery within 28 days of study enrollment (other than diverting colostomy)
  * Crohn's disease or ulcerative colitis requiring hospitalization, surgery or immunosuppressive medications
* Prior allergic reaction to 5-Fluorouracil or oxaliplatin
* Any evidence of distant metastases (M1)
* Extension of malignant disease into the anal canal
* Pregnant as determined by a positive serum pregnancy test within 14 days prior to registration on study (for females of childbearing potential)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2014-12-04 (Actual); Primary Completion 2018-05-14 (Actual); Study Completion 2021-05-13 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity for continuous infusional 5-Fluorouracil given concurrently with short course pelvic radiation | Up to 21 days
  To determine the maximum tolerated dose of continuous infusional 5-Fluorouracil, up to a target dose of 200 mg/m^2/day, given concurrently with short course radiation followed by neoadjuvant FOLFOX chemotherapy and planned surgical resection for locally advanced rectal cancer. Assessed using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.

SECONDARY OUTCOMES:
Pathological response rate for subjects treated with concurrent 5-FU | Up to at least 5 years
  To determine the rates of pathologic response for subjects treated with 5-FU together with neoadjuvant, short course pelvic RT.
Complete response rate with radiographic imaging prior to surgery | Up to 8 weeks after completion of pre-operative chemotherapy
  To determine the rate of complete response prior to surgery.
Three-year rate of local-regional recurrence for all subjects enrolled on the study | 3 years
  To determine the rates of local-regional recurrence for subjects treated with 5-FU together with neoadjuvant, short course pelvic RT.
Adverse events at any time | 30 days after surgery
  To determine the incidence of all toxicity (gastrointestinal and non-gastrointestinal) associated with protocol treatment in the preoperative period, the postoperative period, and therefore assess the tolerability of the combination regimen.
Three-year rate of disease-free survival for all subjects enrolled on the study | 3 years
  To determine the disease-free survival for subjects treated with 5-FU together with neoadjuvant, short course pelvic RT.
Postoperative morbidity rates | Up to 30 days after surgery
Postoperative mortality rates | Up to 30 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Emma C Fields, MD, Principal Investigator — Massey Cancer Center
Locations (1):
- Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia, United States